CLINICAL TRIAL: NCT00456716
Title: A Phase II Trial of Sorafenib in BAC or Never-Smokers With Any Lung Adenocarcinoma
Brief Title: Sorafenib in BAC or Never-Smokers With Lung Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: Bayer (Industry); Amgen (Industry)
Responsible Party: Howard Jack West, M.D., Swedish Medical Center, Swedish Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC 0639
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Lung Cancer
Keywords: BAC lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sorafenib — 400mg po bid
  Other Names: BAY 43-9006

SUMMARY:
Open label study of sorafenib

DETAILED DESCRIPTION:
Open label study using oral sorafenib 800 mg daily in any stage III-IV BAC lung cancer and Stage III-IV adenocarcinoma of the lung in nonsmokers (less than < 100 cigarettes lifetime).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Life expectancy > 12 weeks
* Biopsy-proven BAC or adenocarcinoma
* Willing to provide smoking status
* Selected IIIB or stage IV cancer that is incompletely resected or unresectable

Exclusion Criteria:

* O2 saturation < 88% on room air
* Pregnant or nursing women
* Surgery or radiation therapy within 4 weeks of starting study
* Major heart condition within 6 months of starting therapy
* Certain concomitant medications prohibited

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Response rate | January 2009
One-year survival | January 2009
Median survival | January 2009

SECONDARY OUTCOMES:
Median progression-free survival | January 2009
Toxicities | January 2009

CONTACTS AND LOCATIONS:
Overall Officials: Howard J West, M.D., Principal Investigator — Swedish Cancer Institute
Locations (1):
- Swedish Cancer Institute, Seattle, Washington, United States